CLINICAL TRIAL: NCT02665182
Title: Up-positioning of the Testes as Supportive Therapy in Patients With Acute Orchitis - a Randomized Controlled Trial
Brief Title: Up-positioning of the Testes as Supportive Therapy in Patients With Acute Orchitis
Acronym: EleScro
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SP12-1
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Orchitis; Testicular Diseases
Keywords: orchitis; testicular diseases
MeSH Terms: conditions — Orchitis; Testicular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Up-positioning of the testes (Experimental): Patients receive standard medical therapy and supportive therapy
  Interventions: Behavioral: Up-positioning of the testes
- Medical therapy only (No Intervention): Patients receive standard medical therapy only

INTERVENTIONS:
Behavioral: Up-positioning of the testes — Patients in the experimental arm are asked to elevate their testes during the treatment.
  Arms: Up-positioning of the testes

SUMMARY:
This is a single-blinded RCT evaluating the value of up-positioning of the testes as supportive therapy in patients receiving antimicrobial treatment due to acute bacterial orchitis.

ELIGIBILITY:
Inclusion Criteria:

* acute orchitis confirmed clinically and in scrotal ultrasound
* age >=18 yrs

Exclusion Criteria:

* previous treatment of orchitis,
* need for exploration of the scrotum,
* need for hospitalization,
* physical and mental status not allowing for up-positioning of the testes during treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-07; Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Time to alleviation of symptoms | 10 days
Time to clinical resolution of local symptoms | 10 days

SECONDARY OUTCOMES:
Testicular pain | 10 days
Testicular swelling | 10 days
Testicular erythema | 10 days
Scrotal pain intensity | 10 days
Quality of life | 10 days
Body temperature | 10 days
Heart rate | 10 days
Duration of up-positioning of testes per day | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Sławomir Poletajew, MD PhD, Study Director — Medical University of Warsaw
Locations (1):
- Sławomir Poletajew, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No